CLINICAL TRIAL: NCT02451605
Title: Regional Blockade for Knee Prothesis Surgery: Comparison Between Femoral, Sciatic and Adductor Canal Block
Brief Title: Regional Anesthesia for Knee Prothesis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Pierre Goffin, Clinical assistant, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-000677-39
Record Dates: First submitted 2015-05-12; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Total Knee Replacement
Keywords: surgery
MeSH Terms: interventions — Ropivacaine; Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Femoral nerve blockade (Active Comparator): In this group, patient will benefit of an ultrasound guided femoral nerve blockade with continuous catheter infusion as (initial bolus of 20ml of ropivacaine 0.75% follow with 7ml/hour of ropivacaine 0.2%) as analgesic nerve blockade for total knee replacement surgery.
  Interventions: Drug: Analgesic nerve blockade (Ropivacaine); Procedure: Total knee replacement surgery.
- Adductor canal blockade (Active Comparator): In this group, patient will benefit of an ultrasound guided adductor canal blockade with continuous catheter infusion (initial bolus of 20ml of ropivacaine 0.75% follow with 7ml/hour of ropivacaine 0.2%) as analgesic nerve blockade for for total knee replacement surgery.
  Interventions: Drug: Analgesic nerve blockade (Ropivacaine); Procedure: Total knee replacement surgery.
- Subgluteal sciatic nerve blockade (Active Comparator): In this group, patient will benefit of an ultrasound guided subgluteal sciatic nerve blockade with continuous catheter infusion (initial bolus of 20ml of ropivacaine 0.75% follow with 7ml/hour of ropivacaine 0.2%) as analgesic nerve blockade for total knee replacement surgery.
  Interventions: Drug: Analgesic nerve blockade (Ropivacaine); Procedure: Total knee replacement surgery.

INTERVENTIONS:
Drug: Analgesic nerve blockade (Ropivacaine) — Analgesic nerve blockade (Ropivacaine) for total knee replacement surgery.
  Other Names: Regional anesthesia
Procedure: Total knee replacement surgery. — Total knee replacement surgery.

SUMMARY:
Comparison of the analgesics blocks (femoral, adductor canal and sciatic subgluteal nerve) for total replacement knee surgery.

DETAILED DESCRIPTION:
Adductor canal block shows a beneficial effect for knee surgery. Mainly because he prevent for muscular weakness; adverse effect meet with femoral block and delaying the early active mobilization.

The investigators want to compare the efficacy and safety of this block compared to the femoral and sciatic block.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total knee replacement surgery.

Exclusion Criteria:

* refusal to study,
* coagulation disorder,
* infection at the puncture site,
* preexisting neuropathy,
* allergy to local anesthetics,
* renal or hepatocellular insufficiency,
* context of chronic pain,
* drugs abuse,
* pregnant patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pain measurement with numeric pain scale : from 0 to 10 (maximal pain) in rest condition | up to day 7
  Pain assessment and evolution in postoperative period (passive condition)
Pain measurement with numeric pain scale (from 0 to 10) during active motorized mobilization (Kinetic) | up to day 7
  Pain assessment and evolution in postoperative period (active condition)

SECONDARY OUTCOMES:
Postintervention nausea vomiting | at hour 0, at hours 6, at day 1
  question : present or not
Patient satisfaction | at day 1
  Questionnaire of patient felling and satisfaction. Choice within gradual felling : bad, middle, good, excellent
Opioid consumption | up to 48 hours
  doses of piritramid (synthetic opioid) administrated with patient control rescue analgesia device.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Brichant, Study Chair — University of Liege
Locations (1):
- University og Liege, University Hospital, Liège, Belgium